CLINICAL TRIAL: NCT06850714
Title: Evaluation of the Use of Bifidobacterium Breve PRL2020 in Preventing Side Effects From Amoxicillin or Amoxicillin/Clavulanic Acid Antibiotic Use: A Randomized Controlled Trial
Brief Title: Evaluation of Bifidobacterium Breve PRL2020 in Preventing Antibiotic-Associated Side Effects From Amoxicillin or Amoxicillin/Clavulanic Acid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CESU/77/06.09.2023
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Antibiotic Side Effect
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic + Antibiotic Group (Probiotic Group) (Experimental): Participants in this group will receive Amoxicillin or Amoxicillin/Clavulanic Acid as prescribed by their physician, and a probiotic as add-on for the duration of antibiotic therapy (6-10 days).
  Interventions: Dietary Supplement: Bifidobacterium breve PRL2020 (Brevicillin®); Drug: Amoxicillin or Amoxicillin/Clavulanic Acid
- Antibiotic-Only Group (Control Group) (Active Comparator): Participants in this group will receive only Amoxicillin or Amoxicillin/Clavulanic Acid as per medical prescription.
  Interventions: Drug: Amoxicillin or Amoxicillin/Clavulanic Acid

INTERVENTIONS:
Dietary Supplement: Bifidobacterium breve PRL2020 (Brevicillin®) — Probiotic Bifidobacterium breve PRL2020 (Brevicillin®) at a dose of 20 billion CFU per day (one stick in the morning and one in the evening).
  Other Names: Brevicillin®, PharmExtracta S.p.A.
  Arms: Probiotic + Antibiotic Group (Probiotic Group)
Drug: Amoxicillin or Amoxicillin/Clavulanic Acid — Treatment of Amoxicillin or Amoxicillin/Clavulanic Acid as per medical prescription.

SUMMARY:
This study aims to evaluate the efficacy and safety of the probiotic Bifidobacterium breve PRL2020 in preventing gastrointestinal and extra-intestinal side effects caused by Amoxicillin or Amoxicillin/Clavulanic Acid in pediatric patients. The study will compare a treatment group receiving the probiotic alongside antibiotics with a control group receiving antibiotics alone. The primary focus is on reducing antibiotic-induced intestinal discomfort through microbiota modulation.

DETAILED DESCRIPTION:
Antibiotic therapy, particularly with Amoxicillin and Amoxicillin/Clavulanic Acid, is widely used to treat bacterial infections in children. However, these antibiotics often disrupt the gut microbiota, leading to gastrointestinal side effects such as diarrhea, bloating, abdominal pain, and constipation. This imbalance can reduce the abundance of beneficial bacterial species, including bifidobacteria, potentially leading to long-term gastrointestinal dysbiosis.

This observational, non-profit study aims to evaluate the efficacy and safety of Bifidobacterium breve PRL2020 (Brevicillin®), a probiotic strain with demonstrated resistance to Amoxicillin and Amoxicillin/Clavulanic Acid. Prior research has shown that this strain has a high minimum inhibitory concentration (MIC) of 32-64 μg/mL, making it a promising candidate for preventing antibiotic-associated gut microbiota alterations.

The study will recruit 800 pediatric patients (ages 3-12 years) who require antibiotic therapy for infections. Participants will be randomized into two groups:

Probiotic Group: Receives Bifidobacterium breve PRL2020 (20 billion CFU per day) alongside antibiotic treatment.

Control Group: Receives antibiotics only, without probiotic supplementation. The primary outcome will be the evaluation of gastrointestinal symptoms and stool consistency using the Bristol Stool Scale and a VAS symptom scale (0-7 points) over a 15-day period (treatment duration + follow-up). The secondary outcome will assess the safety and tolerability of the probiotic intervention.

Clinical data will be collected via a daily symptom diary maintained by caregivers, including frequency of bowel movements, stool quality, presence of abdominal pain, and other potential side effects. Statistical analysis will determine whether Bifidobacterium breve PRL2020 significantly reduces antibiotic-associated gastrointestinal disturbances compared to the control group.

This study is expected to provide critical insights into the role of probiotic supplementation in mitigating antibiotic-induced dysbiosis, potentially shaping future guidelines for pediatric antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 12 years
* Requiring antibiotic therapy with Amoxicillin or Amoxicillin/Clavulanic Acid
* Ability to comply with the study protocol (parents/caregivers must complete symptom diaries)

Exclusion Criteria:

* Use of any antibiotic therapy within 3 months before study enrollment
* Known gastrointestinal diseases (e.g., inflammatory bowel disease, celiac disease)
* History of chronic diarrhea or constipation
* Allergy to probiotics or study interventions
* Any immunocompromised state

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2025-02-23 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Antibiotic-Associated Gastrointestinal Symptoms | 15 days (treatment duration + follow-up)
  Evaluation of changes in gastrointestinal symptoms (diarrhea, bloating, abdominal pain, constipation) using the Bristol Stool Scale and a VAS symptom scale (0-7 points). Participants will document symptoms in a daily symptom diary. A significant reduction in symptoms in the probiotic group compared to the control group will indicate efficacy.

SECONDARY OUTCOMES:
Safety and Tolerability of Bifidobacterium breve PRL2020 | 15 days
  Assessment of adverse events or intolerance to the probiotic supplementation.
Incidence of Antibiotic-Associated Diarrhea (AAD) | 15 days
  Proportion of participants developing diarrhea (≥3 loose stools/day for ≥2 days) as per WHO definition.
Changes in Stool Consistency and Frequency | 15 days
  Stool consistency will be assessed using the Bristol Stool Form Scale (BSFS), a validated 7-point scale where:
  Score 1 = Separate hard lumps (severe constipation), Score 7 = Watery, entirely liquid stools (severe diarrhea). Higher scores indicate looser stool consistency and a worse outcome in cases of diarrhea. Lower scores indicate constipation.
  Stool frequency will be recorded as the number of bowel movements per day.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine & Technological Innovation Dept. University of Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartlett JG. Clinical practice. Antibiotic-associated diarrhea. N Engl J Med. 2002 Jan 31;346(5):334-9. doi: 10.1056/NEJMcp011603. No abstract available. PMID 11821511
- [Background] Salvo F, Polimeni G, Moretti U, Conforti A, Leone R, Leoni O, Motola D, Dusi G, Caputi AP. Adverse drug reactions related to amoxicillin alone and in association with clavulanic acid: data from spontaneous reporting in Italy. J Antimicrob Chemother. 2007 Jul;60(1):121-6. doi: 10.1093/jac/dkm111. Epub 2007 Apr 21. PMID 17449881
- [Background] Caron F, Ducrotte P, Lerebours E, Colin R, Humbert G, Denis P. Effects of amoxicillin-clavulanate combination on the motility of the small intestine in human beings. Antimicrob Agents Chemother. 1991 Jun;35(6):1085-8. doi: 10.1128/AAC.35.6.1085. PMID 1929247
- [Background] Yang L, Bajinka O, Jarju PO, Tan Y, Taal AM, Ozdemir G. The varying effects of antibiotics on gut microbiota. AMB Express. 2021 Aug 16;11(1):116. doi: 10.1186/s13568-021-01274-w. PMID 34398323
- [Background] Mancabelli L, Mancino W, Lugli GA, Argentini C, Longhi G, Milani C, Viappiani A, Anzalone R, Bernasconi S, van Sinderen D, Ventura M, Turroni F. Amoxicillin-Clavulanic Acid Resistance in the Genus Bifidobacterium. Appl Environ Microbiol. 2021 Mar 11;87(7):e03137-20. doi: 10.1128/AEM.03137-20. Print 2021 Mar 11. PMID 33483308
- [Background] Di Pierro F, Campedelli I, De Marta P, Fracchetti F, Del Casale A, Cavecchia I, Matera M, Cazzaniga M, Bertuccioli A, Guasti L, Zerbinati N. Bifidobacterium breve PRL2020: Antibiotic-Resistant Profile and Genomic Detection of Antibiotic Resistance Determinants. Microorganisms. 2023 Jun 24;11(7):1649. doi: 10.3390/microorganisms11071649. PMID 37512822